CLINICAL TRIAL: NCT01900769
Title: Calculating Blood Volume by Dilution of Hemoglobin - Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kai Schoenhage (Other)
Responsible Party: Sponsor-Investigator, Kai Schoenhage, Assistant Professor, Anesthesiology Director of Perioperative Services, Director of Liver Transplant Anesthesia, Department of Anesthesiology, University of Arizona
Organization: University of Arizona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-0077
Record Dates: First submitted 2013-07-12; First posted 2013-07-16 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Determine Validity of Concept of Using Hemoglobin Dilution to Assess/Measure Blood Volume.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood Volume Dilution (Experimental)
  Interventions: Drug: Blood Volume Dilution

INTERVENTIONS:
Drug: Blood Volume Dilution

SUMMARY:
Although blood volume is such an important parameter in everyday clinical medicine it cannot be measured easily. As a matter of fact, it is almost never measured but estimated or calculated based upon numbers derived from mostly healthy patients.

The investigators do not even know whether someone's normal - i.e. before a surgery - blood volume is actually anywhere close to the generally accepted estimate or calculation.

Tests exist in which a substance of known concentration is diluted in a person's blood volume and the resulting concentration is then measured, which allows the blood volume to be calculated. However, none of these tests can be completed at the bedside since they are not fast and require considerable set-up.

This study turns the above approach upside-down: we will dilute the blood slightly with a known small volume of an intravenous fluid commonly used in many clinical settings and measure the concentra-tion of hemoglobin - the oxygen carrier contained in red blood cells - before and after adding the fluid. That allows for similar calculations without using neither specialized substances nor equipment.

Hemoglobin is routinely measured in laboratories and is often a routine test before and during surg-eries and in intensive care units.

Devices that can measure hemoglobin through the skin without actually drawing any blood are avail-able. If found comparable to laboratory determination of hemoglobin they could provide for a bedside and almost real-time assessment of blood volume, something that could be extremely valuable for de-cision making in critical areas of medicine and promoting goal directed therapies.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults of normal constitution (weight/height)

Exclusion Criteria:

* any ongoing or recent infusions (< 24h ago) of any fluid/substance
* morbid obesity
* heart disease
* hypertension
* coagulopathy (bleeding disorder)
* therapy with anti- or procoagulants
* transfusion of any blood product
* therapy with diuretics
* therapy with vasopressors
* vasodilators or inotropes
* acute or chronic infections
* immunocompromised status
* hemodynamically unstable
* hemorrhage (bleeding)
* recent surgery
* pregnancy
* younger than 18 years old

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
matching BV by Hemoglobin dilution (lab) | 5 - 40 minutes

SECONDARY OUTCOMES:
matching BV by Hemoglobin dilution (SpHb) | 5 - 40 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Kai Schoenhage, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Medical Center, Tucson, Arizona, United States